CLINICAL TRIAL: NCT04392011
Title: Assessing the Pharmacokinetics and Drug Interaction Liability of Kratom, an Opioid-like Natural Product
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mary Paine, Professor, Washington State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 17823; U54AT008909 (NIH)
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Results first posted 2023-06-08 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Interaction Drug Food
Keywords: Pharmacokinetics; Kratom; Mitragynine; Midazolam; Dextromethorphan; Natural product
MeSH Terms: interventions — Midazolam; Dextromethorphan; mitragynine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Six non-naive* subjects (3 males, 3 females) will be administered a single low dose of a well-characterized kratom product (2 g) by mouth as a tea. These subjects may or may not choose to participate in Arms 2a and 2b. For subjects who will participate in Arms 2a and 2b, a washout period of 7 days will separate Arm 1 and Arm 2. Plasma will be collected from 0-120 hours and during the washout period. Urine will be collected from 0-120 hours.
  *Non-naive subjects are defined as intermittent users who consume 2-8 g kratom at least once per month but no more than three times daily within the last six months prior to screening and are willing to abstain for several weeks.
  Interventions: Dietary Supplement: Kratom
- Arm 2 (Experimental): Arm 2 is divided into Arms 2a and 2b. Twelve non-naive subjects (6 males, 6 females) will participate in Arm 2a. Subjects who participate in this study arm will be administered an oral probe drug cocktail of dextromethorphan HBr (2 x 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma will be collected from 0-24 hours. Urine will be collected from 0-24 hours. A washout period of 7 days will separate Arms 2a and 2b.
  For Arm 2b, the same 12 subjects will be administered a combination of a well-characterized kratom product (2 g) by mouth as a tea with an oral probe drug cocktail consisting of dextromethorphan HBr (2, 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma will be collected from 0-12 hours and during a midpoint collection within 5 days of the 24-hour blood collection. Urine will be collected from 0-24 hours.
  Interventions: Drug: Midazolam HCl; Drug: Dextromethorphan HBr; Dietary Supplement: Kratom

INTERVENTIONS:
Drug: Midazolam HCl — Oral syrup, 2 mg/mL
  Arms: Arm 2
Drug: Dextromethorphan HBr — Oral liquid capsules, 15 mg
  Arms: Arm 2
Dietary Supplement: Kratom — Kratom (Moon Kratom Yellow Indonesian, lot 51) is supplied as a dry leaf powder in clear plastic bags, each weighing 5 kg. Two g of kratom dry leaf powder will be stirred into 240 mL of hot water to make a tea. The tea will be cooled to 50 degrees Celsius before administration. Subjects will drink the tea within 10 minutes of administration.

SUMMARY:
Kratom is a botanical natural product that has opioid-like effects. Kratom is commonly used to self-treat withdrawal symptoms associated with opioid addiction, as well as pain. Kratom products include pills, extracts, and powders, most of which contain two primary psychoactive constituents: mitragynine and 7-hydroxymitragynine. Preliminary data from the investigator's laboratory has shown that these two constituents and extracts made from commercially available kratom products are strong inhibitors of the drug metabolizing enzymes cytochrome P450 (CYP) 2D6 and CYP3A4. These enzymes are responsible for metabolizing more than 50% of marketed drugs, including several opioids, benzodiazepines, and antidepressants. Thus, co-consumption of kratom products with drugs metabolized by CYP2D6 and CYP3A4 could increase the risk of serious adverse effects. The effects of a well-characterized kratom product on CYP2D6 and CYP3A4 activity will be assessed in healthy volunteers using a 'cocktail' approach consisting of the validated probe drugs dextromethorphan and midazolam. Results will (1) provide useful information regarding risks associated with co-consuming kratom with opioids and other CYP2D6 and CYP3A4 drug substrates and (2) inform the design of future kratom-drug interactions studies.

DETAILED DESCRIPTION:
Many patient groups often supplement their drug regimens with herbal and other natural products (NPs), raising concern for adverse NP-drug interactions. Due to a lack of rigorous guidelines for assessing the risk of NP-drug interactions, the NIH-funded Center of Excellence for Natural Product-Drug Interaction Research (NaPDI Center) was established to facilitate the identification, evaluation, and dissemination of potentially clinically relevant pharmacokinetic NP-drug interactions.Kratom is one of four high priority NPs selected by the NaPDI Center for rigorous study of drug interaction potential.

Kratom (Mitragyna speciosa) is a tree native to Southeast Asia that produces constituents with opioid-like effects. Oral supplements made from the leaves are readily available in the United States and are used for several purported medicinal benefits, such as pain relief, treatment of post-traumatic stress disorder, and management of opioid addiction. Two psychoactive constituents of the kratom leaf, mitragynine and 7- hydroxymitragynine, are believed to contribute to these effects.

Calls to poison control centers in the United States involving kratom exposures increased from 2011 to 2017 by 52-fold. More than one-third of the calls reported combined use of kratom with other substances, including opioids and benzodiazepines. In October 2017, the opioid crisis was declared a public health emergency. Many opioids are metabolized by the major drug metabolizing enzymes CYP2D6 and CYP3A4, which have been shown to be inhibited by an extract prepared from a well-characterized kratom product and purified major kratom constituents, including mitragynine and 7-hydroxymitragynine. As such, co-consuming kratom with these opioids could increase the risk of serious adverse effects via inhibition of opioid metabolism, notably respiratory depression, the primary cause of death from opioid overdose.

The purpose of this study is to assess the effects of a well-characterized kratom product on CYP2D6 and CYP3A4 activity in healthy volunteers using a cocktail approach consisting of the validated probe drugs dextromethorphan and midazolam. The primary objective is to evaluate the potential for a pharmacokinetic kratom-drug interaction with midazolam, a 'probe' drug for CYP3A4, when administered to participants previously exposed to kratom. Secondary objectives are to evaluate the pharmacokinetics of kratom constituents and the effect of kratom on the pharmacokinetics of dextromethorphan, a probe drug for CYP2D6.

Results will be used to develop physiologically-based pharmacokinetic (PBPK) models to predict the likelihood and magnitude of kratom-drug interactions, including those involving opioids. These PBPK models could be adapted to other CYP2D6 and CYP3A4 drug substrates with high abuse potential (e.g., benzodiazepines and 'Z-drugs') and used to inform the design of future kratom-drug interactions studies.

ELIGIBILITY:
Inclusion Criteria:

* Not taking any medications (prescription and non-prescription) or dietary/herbal supplements known to alter the pharmacokinetics of either study drug or kratom constituents
* Willing to abstain from consuming dietary/herbal supplements, including kratom, and citrus juices for several weeks
* Willing to abstain from consuming caffeinated beverages or other caffeine-containing products the evening before and morning of the first day of a study arm
* Willing to abstain from consuming any alcoholic beverages for one day prior to any study day, during the 14-hour inpatient days, and for the 5 and/or 1 outpatient visit(s) following 14-hour visit
* Willing to use an acceptable method of contraception that does not include oral contraceptive pills or patches (such as abstinence, copper IUD, condom)
* Have the time to participate
* Are non-naïve kratom users (intermittent users who are not trying to quit but willing to abstain for several weeks)
* Carry a CYP2D6 genotype designated as having an intermediate, extensive, or ultra-extensive metabolizer phenotype
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for the subject to comply with the requirements of the study

Exclusion Criteria:

* Men and women under the age of 18 or over the age of 55
* Unwilling to abstain from kratom for several weeks
* Any current major illness or chronic illness such as (but not limited to) kidney disease, hepatic disease, diabetes mellitus, hypertension, coronary artery disease, chronic obstructive pulmonary disease, cancer, or HIV/AIDS
* History of anemia or any other significant hematologic disorder
* History of drug or alcohol addiction or major psychiatric illness
* A need for chronic opioid analgesics
* Use of opioid analgesics 3 weeks prior to initiation of the study
* An imminent likely need for opioid analgesics (e.g., planned dental or surgical procedure)
* Female and pregnant or nursing
* Have a history of allergy to dextromethorphan, midazolam, or related drugs
* Have a history of intolerance or allergy to kratom or opioids
* Taking concomitant medications, both prescription and non-prescription (including dietary supplements/herbal products), known to alter the pharmacokinetics of either study drug or kratom constituents
* Carry a CYP2D6 genotype designated as having a poor metabolizer phenotype
* Presence of a condition or abnormality that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Washington State University College of Pharmacy and Pharmaceutical Sciences, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Post S, Spiller HA, Chounthirath T, Smith GA. Kratom exposures reported to United States poison control centers: 2011-2017. Clin Toxicol (Phila). 2019 Oct;57(10):847-854. doi: 10.1080/15563650.2019.1569236. Epub 2019 Feb 20. PMID 30786220

RESULTS

PARTICIPANT FLOW:
Groups:
- Kratom Only(1 Day)-Washout(7 Days)-Drug Cocktail(1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day): Six non-naive* subjects (3 males, 3 females) were administered a single low dose of a well-characterized kratom product (2 g) by mouth as a tea. Plasma and urine were collected from 0-120 hours. Subjects then underwent a washout period of at least 7 days before continuing the study. The same six subjects were then administered an oral probe drug cocktail of dextromethorphan HBr (2 x 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma and urine were collected from 0-24 hours. Subjects then underwent a washout period of at least 7 days.
  The same 6 subjects were then administered kratom (2 g) with an oral probe drug cocktail consisting of dextromethorphan HBr (2, 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma was collected from 0-12 hours and during a midpoint collection within 5 days of the 24-hour blood collection. Urine was collected from 0-24 hours.
  *Non-naive subjects are defined as intermittent users who consume 2-8 g kratom at least once per month but no more than three times daily within the last six months prior to screening and are willing to abstain for several weeks.
- Drug Cocktail (1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day): Seven non-naive* subjects (4 males and 3 females) were administered an oral probe drug cocktail of dextromethorphan HBr (2 x 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma and urine were collected from 0-24 hours. Subjects then underwent a washout period of at least 7 days.
  Six of those subjects were then administered kratom (2 g) with an oral probe drug cocktail consisting of dextromethorphan HBr (2, 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma was collected from 0-12 hours and during a midpoint collection within 5 days of the 24-hour blood collection. Urine was collected from 0-24 hours.
  *Non-naive subjects are defined as intermittent users who consume 2-8 g kratom at least once per month but no more than three times daily within the last six months prior to screening and are willing to abstain for several weeks.
Period: Kratom Only
Arm/Group | Kratom Only(1 Day)-Washout(7 Days)-Drug Cocktail(1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day) | Drug Cocktail (1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day)
Started | 8 | 0
Completed | 6 | 0
Not Completed | 2 | 0
Period: Washout
Arm/Group | Kratom Only(1 Day)-Washout(7 Days)-Drug Cocktail(1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day) | Drug Cocktail (1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day)
Started | 6 | 0
Completed | 6 | 0
Not Completed | 0 | 0
Period: Drug Cocktail Only
Arm/Group | Kratom Only(1 Day)-Washout(7 Days)-Drug Cocktail(1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day) | Drug Cocktail (1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day)
Started | 6 | 7
Completed | 6 | 7
Not Completed | 0 | 0
Period: Washout
Arm/Group | Kratom Only(1 Day)-Washout(7 Days)-Drug Cocktail(1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day) | Drug Cocktail (1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day)
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1
Period: Kratom + Drug Cocktail
Arm/Group | Kratom Only(1 Day)-Washout(7 Days)-Drug Cocktail(1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day) | Drug Cocktail (1 Day)-Washout(7 Days)-Kratom+Drug Cocktail(1 Day)
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Kratom Alone - Washout - Drug Cocktail - Washout - Kratom+Drug Cocktail: Six non-naive* subjects (3 males, 3 females) were administered a single low dose of a well-characterized kratom product (2 g) by mouth as a tea. Plasma will be collected from 0-120 hours and during the washout period. Urine was collected from 0-120 hours. After a washout of at least 7 days, the subjects were then administered an oral probe drug cocktail of dextromethorphan HBr (2 x 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma and urine were collected from 0-24 hours. After a washout period of at least 7 days, they were then administered a combination of a well-characterized kratom product (2 g) by mouth as a tea with an oral probe drug cocktail consisting of dextromethorphan HBr (2, 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma was collected from 0-12 hours and during a midpoint collection within 5 days of the 24-hour blood collection. Urine was collected from 0-24 hours.
- Drug Cocktail - Washout - Kratom+Drug Cocktail: Seven non-naive* subjects (4 males, 3 females) were administered an oral probe drug cocktail of dextromethorphan HBr (2 x 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma and urine were collected from 0-24 hours. After a washout period of at least 7 days, they were then administered a combination of a well-characterized kratom product (2 g) by mouth as a tea with an oral probe drug cocktail consisting of dextromethorphan HBr (2, 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma was collected from 0-12 hours and during a midpoint collection within 5 days of the 24-hour blood collection. Urine was collected from 0-24 hours.
- Total: Total of all reporting groups
Arm/Group | Kratom Alone - Washout - Drug Cocktail - Washout - Kratom+Drug Cocktail | Drug Cocktail - Washout - Kratom+Drug Cocktail | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 6 | 10
  Asian | 2 | 1 | 3
  Black | 1 | 0 | 1
  More than 1 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Midazolam Area Under the Concentration vs. Time Curve (AUC)
Description: Area under the plasma concentration time curve (AUC) of midazolam
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, 24, 48, 72 , 96, 120, and 144 hours
Population: Although 13 subjects completed the drug cocktail arm, only the 12 subjects that completed both that and the kratom + drug cocktail arm were analyzed, as the drug cocktail arm was intended as a baseline to which the kratom + drug cocktail arm would be compared.
Measure: Geometric Mean (90% Confidence Interval); unit: nM * hr
Groups:
- Drug Cocktail: Thirteen subjects were administered an oral probe drug cocktail consisting of dextromethorphan HBr (2, 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma was collected from 0-12 hours and during a midpoint collection within 5 days of the 24-hour blood collection. Urine was collected from 0-24 hours.
- Kratom + Drug Cocktail: Twelve subjects were administered kratom (2 g) with an oral probe drug cocktail consisting of dextromethorphan HBr (2, 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma was collected from 0-12 hours and during a midpoint collection within 5 days of the 24-hour blood collection. Urine was collected from 0-24 hours.
Arm/Group | Drug Cocktail | Kratom + Drug Cocktail
Number analyzed (Participants) | 12 | 12
nM * hr | 58.3 [48.5 to 70.2] | 80.8 [64.2 to 102]
Statistical Analysis 1: Comparison: Drug Cocktail vs Kratom + Drug Cocktail; Test type: Other; AUC ratio (geometric mean) = 1.39, 90% CI 2-sided [1.23 to 1.57]

2. Secondary Outcome: Dextromethorphan Area Under the Concentration vs. Time Curve (AUC)
Description: Area under the plasma concentration time curve (AUC) of dextromethorphan
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, 24, 48, 72, 96, 120, and 144 hours
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: nM*h
Arm/Group | Drug Cocktail | Kratom + Drug Cocktail
Number analyzed (Participants) | 12 | 12
nM*h | 46.5 [19.4 to 112] | 46.2 [19.2 to 112]
Statistical Analysis 1: Comparison: Drug Cocktail vs Kratom + Drug Cocktail; Test type: Other; AUC ratio (geometric mean) = 0.99, 90% CI 2-sided [0.83 to 1.19]

3. Secondary Outcome: Mitragynine Area Under the Concentration vs. Time Curve (AUC)
Description: Area under the concentration vs. time curve (AUC) of mitragynine.
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, 24, 48, 72, 96, and 120 hours
Measure: Median (Full Range); unit: nM x h
Groups:
- Kratom Alone: Six non-naive* subjects were administered a single low dose of a well-characterized kratom product (2 g) by mouth as a tea. Plasma and urine were collected from 0-120 hours. Subjects then underwent a washout period of at least 7 days before continuing the study.
Arm/Group | Kratom Alone
Number analyzed (Participants) | 6
nM x h | 388 [300 to 1240]

4. Secondary Outcome: Midazolam and Dextromethorphan Cmax
Description: Maximum concentration (Cmax) of midazolam and dextromethorphan
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, 24, 48, 72, 96,120, and 144 hours
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: nM
Groups:
- Drug Cocktail: Thirteen subjects were administered an oral probe drug cocktail of dextromethorphan HBr (2 x 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma and urine were collected from 0-24 hours. Subjects then underwent a washout period of at least 7 days.
Arm/Group | Drug Cocktail | Kratom + Drug Cocktail
Number analyzed (Participants) | 12 | 12
nM
  midazolam | 21.1 [17.2 to 26.0] | 31.6 [26.4 to 38.0]
  dextromethorphan | 4.57 [2.07 to 10.1] | 4.30 [2.06 to 9.28]
Statistical Analysis 1: Comparison: Drug Cocktail vs Kratom + Drug Cocktail; Test type: Other; Cmax ratio (midazolam) = 1.50, 90% CI 2-sided [1.32 to 1.70]
Statistical Analysis 2: Comparison: Drug Cocktail vs Kratom + Drug Cocktail; Test type: Other; Cmax ratio (dextromethorphan) = 0.96, 90% CI 2-sided [0.78 to 1.19]

5. Secondary Outcome: Mitragynine Cmax
Description: Maximum plasma concentration of mitragynine.
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, 24, 48, 72, 96, and 120 hours
Measure: Median (Full Range); unit: nM
Arm/Group | Kratom Alone
Number analyzed (Participants) | 6
nM | 81.9 [50.1 to 177]

6. Secondary Outcome: Midazolam and Dextromethorphan Half-life
Description: Time to reach one-half of the concentration of midazolam and dextromethorphan
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, 24, 48, 72, 96,120, and 144 hours
Population: as for outcome 1
Measure: Geometric Mean (90% Confidence Interval); unit: h
Groups:
- Drug Cocktail: Thirteen subjects were administered an oral probe drug cocktail of dextromethorphan HBr (2 x 15 mg liquid capsules; 30 mg total) and midazolam HCl (1.25 mL of 2 mg/mL syrup; 2.5 mg total). Plasma and urine were collected from 0-24 hours.
Arm/Group | Drug Cocktail | Kratom + Drug Cocktail
Number analyzed (Participants) | 12 | 12
h
  midazolam | 3.85 [3.25 to 4.56] | 4.12 [3.45 to 4.92]
  dextromethorphan | 6.87 [5.85 to 8.06] | 6.84 [5.62 to 8.34]
Statistical Analysis 1: Comparison: Drug Cocktail vs Kratom + Drug Cocktail; Test type: Other; half-life ratio (dextromethorphan) = 1.00, 90% CI 2-sided [0.92 to 1.08]
Statistical Analysis 2: Comparison: Drug Cocktail vs Kratom + Drug Cocktail; Test type: Other; half-life ratio (midazolam) = 1.07, 90% CI 2-sided [0.98 to 1.17]

7. Secondary Outcome: Mitragynine Half Life
Description: Time to reach one-half of the concentration of mitragynine.
Time Frame: 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8,12, 24, 48, 72, 96, and 120 hours
Measure: Median (Full Range); unit: h
Arm/Group | Kratom Alone
Number analyzed (Participants) | 6
h | 45.3 [31.9 to 50.2]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Kratom Alone | Drug Cocktail | Kratom + Drug Cocktail
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 1/8 | 1/13 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kratom Alone (N=8) | Drug Cocktail (N=13) | Kratom + Drug Cocktail (N=12)
headache/lightheadedness (Nervous system disorders) | 1 (3) | 1 (1) | 1 (3)
nausea/vomiting (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT04392011/Prot_SAP_000.pdf
  • Informed Consent Form (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/11/NCT04392011/ICF_001.pdf